CLINICAL TRIAL: NCT05597046
Title: PLANNING PHASE- Qualitative Interviews With Healthcare Professionals to Assist in the Development of a New Patient Reported Outcome Measure (PROM) to Assess Patient's Emotional Wellbeing, and Perceptions of Total Knee Replacement (TKR) Surgery for the Treatment of Knee Arthritis.
Brief Title: Qualitative Interviews With Healthcare Professionals
Status: Completed | Type: Observational
Sponsor: Invibio Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: SYNC01-PP-USA
Record Dates: First submitted 2022-10-25; First posted 2022-10-27 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Total Knee Replacement
Keywords: TKR
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare Professionals: Planning Phase Interviews
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Interviews

SUMMARY:
PLANNING PHASE- Qualitative interviews with Healthcare Professionals to assist in the development of a new Patient Reported Outcome Measure (PROM) to assess patient's emotional wellbeing, and perceptions of Total Knee Replacement (TKR) surgery for the treatment of knee arthritis.

DETAILED DESCRIPTION:
The interviews for the SYNC01-PP-USA project will be conducted in person at the American Association of Hip and Knee Surgeons (AAHKS) annual conference in Dallas, Texas, USA during the 3rd, 4th, and 5th November 2022. The interviews will take approximately 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare Professionals who currently care for patients who have undergone Total Knee Replacement surgery.
* Healthcare Professionals who, in the opinion of the Investigator, can understand the project, co-operate with the interview process and are willing to be interviewed in person.
* Healthcare Professionals who are able to give voluntary, written informed consent to participate in this project and from whom consent has been obtained.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Healthcare Professionals attending the AAKHS conference, Dallas during Thursday 3rd to Saturday 5th November 2022.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
Interview | 30 minutes
  The interview carried out with the HCPs will ascertain their opinions of the issues that patients report after undergoing TKR. The replies (data) collected could be different for each HCP so there is no outcome measure as such for this data. This information collected will be structured around a set number of questions asked in the interview and will be used to form the potential structure and layout of a Patient Reported Outcome Measure (PROM) and to provide background information for the subsequent Phase One of the project which will take place in the UK.

CONTACTS AND LOCATIONS:
Locations (1):
- AAKHS conference, Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided